CLINICAL TRIAL: NCT06829277
Title: Efficacy of Biomimetic Mineralization Approach Plus Soft Laser Irradiation in Management of Dentin Hypersensitivity: A Randomized Clinical Trial
Brief Title: Evaluation of Biomimetic Mineralization Plus Soft Laser Irradiation in Dentin Hypersensitivity Management
Acronym: Rct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Mennatallah Atef Aboulnaga, Lecturer in operative dentistry, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mti-2025-11
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dentin Hypersensitivity
Keywords: Curodont de senz; Laser; Fluoride varnish
MeSH Terms: conditions — Dentin Sensitivity | interventions — Bifluorid 12; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sodium fluoride varnish (Active Comparator): Sodium fluoride varnish
  Interventions: Combination Product: Sodium fluoride varnish
- Curodont De senz (Experimental): Curodont De Senz
  Interventions: Other: Curodont De Senz
- Curodont De Senz plus laser irradiation (Experimental): Curodont De Senz plus laser irradiation
  Interventions: Combination Product: Curodont De Senz plus laser irradiation
- Laser irradiation (Experimental): Laser irradiation
  Interventions: Device: Laser irradiation

INTERVENTIONS:
Combination Product: Sodium fluoride varnish — Sodium fluoride varnish
  Arms: Sodium fluoride varnish
Other: Curodont De Senz — Curodont De Senz
  Arms: Curodont De senz
Combination Product: Curodont De Senz plus laser irradiation — Curodont De Senz plus laser irradiation
  Arms: Curodont De Senz plus laser irradiation
Device: Laser irradiation — Laser irradiation
  Arms: Laser irradiation

SUMMARY:
Randomized clinical trial to investigate the efficacy of diode laser , Biomimetic mineralization desensitizing agents Curodont D'Senz (CS) gel both in combination and alone, and the efficacy of bifluoride 10 (5 % sodium fluoride) varnish alone in cervical dentin hypersensitivity patients. Also, to assess the duration of sensitivity relief immediately after 15 minutes of application, after 2 weeks, after 1 month and 3 months , the null hypothesis that there will be no difference between the treatment groups in different times.

DETAILED DESCRIPTION:
Current research focuses on increasing the mineral density of the dentin surface making it possible to improve its resistance to wear by both acid erosion and abrasion and plugging and sealing open tubules with a calcium and phosphate containing dentin-like substance, which would block diffusion through the tubules into the dentin sub-surface, thereby increasing acid resistance. Self-assembling peptide matrix (P11-4) supplied commercially as Curodont D'Senz (CS) gel (Credentis AG, Windisch, Switzerland) is based on the nanofiber technology that enhances biomimetic repair and the remineralization of dental tissues. Self-assembling peptide matrix hydrogel revealed more reduction of the opened dentinal tubules in comparison to other selected desensitizing toothpaste.lasers have been recently been introduced as another possibility for in-office treatment of DH and may open up new horizons in the treatment of dentin hypersensitivity. Of interest is the fact that the laser irradiation can augment the effect of the desensitizer for a longer duration than when they are used alone. They hypothesized that laser favor the durability of the desensitizer for extended time. Some studies recommend desensitizing agent to remain above tooth surface for one minute before laser irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-60 years old.
* Non-smokers.
* Disease-free patients.
* Good oral hygiene.
* Having at least one teeth suffering from cervical dentin hypersensitivity with VAS pain score ≥5
* Recording pain to thermal, mechanical or tactile stimuli.
* Acceptance to participate in the study

Exclusion criteria:

* Smoking and bad oral hygiene.
* Presence of carious lesions, restorations or fracture in the test area.
* Presence of painful pathology restored less than three months in the test area.
* Using any desen¬sitizing agents.
* Undergo any peri¬odontal surgery in the last 6 months.
* Drug abusers.
* Administration of potent analgesics or anti-inflammatory drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Dentin hypersensitivity | Baseline - 15 minutes- 2 weeks - 1 month - 3 months
  Visual Analogue Scale (VAS) will be used by which 0 is no pain and 10 is severe pain. Pictures are added to the same, as well as colors to guide the patient during selection of pain severity.
  The VAS scale (0-10) is the recommended tool used to evaluate pain of dentin hypersensitivity, and it is the most commonly used in most of the clinical trials. The patient should point out the degree of sensitivity on the VAS scale (0-chart the degree of pain. (VAS >4). A plastic card with figures of facial expressions expressing the degree of pain, color-coded, and numbers guided will be used to ease the process of figuring out the degree of pain. These cards are also useful in standardizing the assessment method for the patient throughout the study and taking records without any verbal or emotional guidance from the assessors.
A- Tactile test | Baseline - 15 minutes- 2 weeks - 1 month - 3 months
  By explorer
B- Evaporative test | Baseline - 15 minutes - 2 weeks- 1 month - 3 months
  By air syringe
C- Thermal Test | Baseline - 15 minutes - 2 weeks- 1 month - 3 months
  By refreigent spray

CONTACTS AND LOCATIONS:
Overall Officials: Aalaa M nabil, Lecturer, Study Chair — MTI University; Ahmed M Sayed, Assis. prof., Study Director — MTI University
Locations (1):
- Mti university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
I will not publish in ICMJE